CLINICAL TRIAL: NCT01629615
Title: A Phase II Trial of BKM120 (a PI3K Inhibitor) in Patients With Triple Negative Metastatic Breast Cancer
Brief Title: A Trial of BKM120 (a PI3K Inhibitor) in Patients With Triple Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Dana-Farber Cancer Institute (Other); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120ZES02T/SOLTI-1103; 2011-006083-45 (EudraCT Number)
Record Dates: First submitted 2012-05-23; First posted 2012-06-27 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; metastatic; triple negative breast cancer; BKM120; SOLTI; PI3K inhibitor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — BKM120 oral capsules. 100 mg daily in cycles of 28 days, until disease progression

SUMMARY:
The purpose of this study is to evaluate the clinical activity of BKM120 in patients with metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, multicenter, single-arm exploratory study of single agent BKM120 in the treatment of metastatic triple negative breast cancer patients.

Patients will first undergo screening, tumor measurement and collection of available tumor block from the primary tumor and/or a metastatic site. Available tumor block is required in all patients per inclusion criteria. Analysis of this tumor block will be used for correlation of predictive markers and clinical response in order to define potential subpopulation that benefit from BKM120.

Following confirmation of eligibility criteria, subjects will be enrolled. BKM120 will then be administered in a 100mg dose, orally, once daily, in a continuous schedule. A treatment cycle is defined as 28 days for the purposes of scheduling procedures and evaluations.

Treatment with BKM120 will continue until disease progression, unacceptable toxicity that precludes any further treatment, and/or discontinuation of the treatment by investigator or patient decision.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and radiologically confirmed metastatic TNBC (Stage IV disease), previously documented by histological analysis, which is ER-negative and PR-negative by IHC and HER2 negative by IHC or FISH/CISH.
* Subjects must have received maximum two prior chemotherapy regimens for metastatic breast cancer.
* Availability of a representative tumor specimen (primary or metastasis, archival tissue or fresh biopsy for patients with biopsiable tumor) at baseline.
* At least one measurable lesion by RECIST 1.1
* Age ≥ 18 years at the day of consenting to the study
* ECOG performance status ≤ 2
* Adequate bone marrow and organ function as defined by the following laboratory values: ANC ≥ 1.0 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9.0 g/dL, INR ≤ 2; serum potassium between 3.0mmol/L and 5.5 mmol/L; Corrected serum calcium between8.0mg/dL and 11.5mg/dL (OR between 1.0mmol/L and 1.5mmol/L of Ionized calcium); serum magnesium between 1.2mg/dL and 3.0 mg/dL; serum creatinine ≤ 1.5 x ULN, ALT and AST within normal range (or ≤ 3.0 x ULN if liver metastases are present); serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome); fasting plasma glucose (FPG) ≤ 140 mg/dL or ≤ 7.8 mmol/L.

Exclusion Criteria:

* Previous treatment with PI3K inhibitors
* Symptomatic CNS metastases
* Patients with controlled and asymptomatic CNS metastases may participate in this trial. As such, the patient must have completed any prior treatment for CNS metastases > 28 days (including radiotherapy and/or surgery) prior to enrollment in this study. Patients with previously treated brain metastases, who are on a stable low dose corticosteroids treatment are eligible
* Concurrent malignancy or malignancy within 3 years of study enrollment (with the exception of adequately treated basal or squamous cell carcinoma or non-melanomatous skin cancer). An exception to this rule are those patients with documented germline mutations in BRCA1 or 2, who may have previous history of cancer
* Any of the following mood disorders as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)

  1. Patients with a history or active episodes of major depression, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, history of suicide attempts or suicidal thoughts (eg. Risk of hurting or harming others) or patients with severe personality disorders (as defined by the DSM-IV) are not eligible. Note: For patients who are treated with psychotropic drugs at baseline, the dose and schedule shall not be changed during the 6 weeks prior to initiation of treatment with the study drug.
  2. ≥ CTCAE v 4.0 grade 3 anxiety
* Patients on concurrent use of other approved or investigational antineoplastic and / or chemotherapy or any continuous or intermittent treatment with therapeutic agents of low molecular weight (excluding monoclonal antibodies) in ≤ 21 days prior to enrollment in this study or who have not recovered from the effects such therapy will not be eligible.
* Radiotherapy ≤ 28 days prior to enrollment in this study or failure to recover from side effects of such therapy at the time of initiation of screening procedures.
* Major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery
* Poorly controlled diabetes mellitus (HbA1c > 8%)
* Active cardiac disease including any of the following:

  1. Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)Note: ECHO/MUGA is only required at baseline if patient has a history of abnormal cardiac test results
  2. QTc > 480 msec on screening ECG (using the QTcF formula
  3. Angina pectoris that requires the use of anti-anginal medication
  4. Ventricular arrhythmias except for benign premature ventricular contractions
  5. Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  6. Conduction abnormality requiring a pacemaker
  7. Valvular disease with documented compromise in cardiac function
  8. Symptomatic pericarditis
* History of cardiac dysfunction including any of the following;

  1. Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  2. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  3. Documented cardiomyopathy
* Treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Chronic treatment with steroids or another immunosuppressive agent. Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed. Patients with previously treated brain metastases, who are on a stable low dose corticosteroids treatment (e.g., dexamethasone 2 mg/day, prednisone 10 mg/day) for at least 14 days before start of study treatment, are eligible
* Other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study (e.g., chronic pancreatitis, active chronic hepatitis etc.)
* History of non-compliance to medical regimen
* Current treatment with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Known history of HIV (testing not mandatory) infection
* Pregnant or nursing (lactating) woman
* Woman of child-bearing potential unwilling to observe total sexual abstinence or to use a double barrier method for birth control throughout the trial. Reliable contraception should be maintained throughout the study and for 6 months after study drug discontinuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Baselga, MD, Study Chair — Massachusetts General Hospital; Eric Winer, MD, Study Chair — Dana-Farber Cancer Institute; Jordi Rodon, MD, Principal Investigator — Hospital Universitario Vall d´Hebron
Locations (7):
- United States (3):
  - Dana-Farber at Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Spain (4):
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Background] Saura C, Lin N, Ciruelos E, Lluch A, Gavilá J, Winer E, Baselga J, Rodón J. A phase II, non-randomized, multicenter, exploratory trial of single agent BKM120 in patients with triple-negative metastatic breast cancer. Poster session presented at: 35th Annual San Antonio Breast Cancer Symposium (SABCS); 2012 December 4th-8th; San Antonio, Texas, United States.
- [Derived] Garrido-Castro AC, Saura C, Barroso-Sousa R, Guo H, Ciruelos E, Bermejo B, Gavila J, Serra V, Prat A, Pare L, Celiz P, Villagrasa P, Li Y, Savoie J, Xu Z, Arteaga CL, Krop IE, Solit DB, Mills GB, Cantley LC, Winer EP, Lin NU, Rodon J. Phase 2 study of buparlisib (BKM120), a pan-class I PI3K inhibitor, in patients with metastatic triple-negative breast cancer. Breast Cancer Res. 2020 Nov 2;22(1):120. doi: 10.1186/s13058-020-01354-y. PMID 33138866
- See also: SOLTI Breast Cancer Research Group — http://www.gruposolti.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BKM120
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population was all recruited population that receives the study treatment
Arm/Group | BKM120
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 53 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
  Spain | 23

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Benefit
Description: Clinical benefit rate (CBR) was defined as the percentage of participants achieving complete response (CR), partial response (PR), or stable disease (SD) for 4 months or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is the complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment then every 3 months up to 2 years. Participants in this study cohort were followed for response on average approximately 2 months.
Population: Intent-to-treat population was all recruited population that receives the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | BKM120
Number analyzed (Participants) | 50
Participants
  Complete response | 0
  Partial response | 0
  Stable disease > 4 months | 6
  Stable disease < 4 months | 11
  Progressive disease | 20
  No evaluable | 13

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) based on the Kaplan-Meier (KM) method is defined as the duration of time from study entry to documented disease progression (PD) or death. Participants alive without PD are censored at the date of last disease assessment. Per RECIST 1.1 criteria: PD is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment then every 3 months up to 2 years. Participants in this study cohort were followed for PFS on average approximately 2 months.
Population: Progression-free survival was analyzed in the intent-to-treat population, defined as all recruited population that receives the study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120
Number analyzed (Participants) | 50
Months | 1.8 [1.6 to 2.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of study enrollment until death from any cause.
Time Frame: 2 years
Population: Overall survival was analyzed in the Intent-to-treat population, defined as all recruited population that receives the study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120
Number analyzed (Participants) | 50
Months | 11.2 [6.2 to 25]

4. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per Common Toxicity Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Adverse events (AEs) were assessed every 2 weeks for the first 2 cycles and every cycle thereafter. Participants were followed for AEs on average approximately 2 months.
Population: The safety population was defined as all the patients who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BKM120
Number analyzed (Participants) | 50
Participants
  Serious Adverse events | 17
  Other Adverse events | 44

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed every 2 weeks for the first 2 cycles and every cycle thereafter. Participants in this study cohort were followed for AEs on average approximately 2 months.
Description: Safety assessments consisted of monitoring by investigators and recording all adverse events, serious adverse events, and the regular monitoring of laboratory evaluations, physical examination, weight, vital signs, and ECG.
  Adverse events were assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | BKM120
All-Cause Mortality (participants affected / at risk) | 29/50
Serious Adverse Events (participants affected / at risk) | 17/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=50)
Fatigue (General disorders) | 4
Papulopustular rash (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Alkalosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Nervous system disorders - Other (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=50)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Watering eyes (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 9
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 16
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 24
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 6
Weight loss (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 5
Libido increased (Psychiatric disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 7
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No